CLINICAL TRIAL: NCT00260910
Title: Progression Evaluation and Genetic Determinants of Hypertension in Chinese - A Follow-up Study of Taiwan SAPPHIRe
Status: Completed | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Tri-Service General Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EC9003003
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2009-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Plasma, serum, urine, and buffy coat
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the progression evaluation and genetic determinations of hypertension in Chinese

DETAILED DESCRIPTION:
Blood pressure is a quantitative trait affected by both genetic and environmental factors. It is known that human essential hypertension does not follow a simple Mendelian mode of inheritance. Stanford-Asian Pacific Program in Hypertension and Insulin Resistance (SAPPHIRe) is an international genetic study, which intends to map the major genetic loci underlying hypertension in sibpairs of Asian-Pacific Chinese and Japanese origin. Based on the data generated through year 1 to year 5, preliminary analysis has not shown positive results in the linkage analysis of genome wide scan data, although association studies of some candidate genes give promising results.

Success in genetic studies may depend on many factors including the selection of the patient population, the identification of intermediate phenotypes, the disease subsets, and the genetic strategy and methodologies employed. According to our previous analysis, presented in SAPPHIRe Steering Committee meetings (twice a year), there is heterogeneity among Chinese and Japanese origins.

In order to reduce heterogeneity of the genetic and environmental background, we will focus our investigation on the Chinese population. Furthermore, besides the variables associated with insulin resistance, which were collected and studied in year 1 through 5 of SAPPHIRe, some more variables will be collected and studied in order to identify most sensible intermediate phenotypes and more homogeneous disease subsets.

Our general approach is to continue analyzing candidate genes as well as perform a complete genome search based on the exiting genome-wide scan data together with old and new phenotype variables.

ELIGIBILITY:
Inclusion Criteria:

* Age of subjects when recruited must be between 35 and 60 years. Subjects over age 60 may also be eligible provided that documentation of their hypertension status prior to age 60 is available.
* Chinese ancestry, i.e. all four grandparents Chinese. Hypertension is defined as follows: systolic BP (SBP) greater than or equal to (>=) 160 mm Hg or diastolic BP (DBP) >= 95 mm Hg or taking 2 medications for high blood pressure (Stage II hypertension). Alternatively the subject could have uncontrolled hypertension, i.e. taking 1 medication for high blood pressure and has either systolic BP >= 140 or diastolic >= 90 mm Hg.

Exclusion Criteria:

* One of the affected sibs is adopted (i.e. no parent in common) or if the sibs have only one parent in common.
* Both parents have been treated for hypertension before the age of 60. If offspring reports about their parents' hypertension status are conflicting, then a single reliable report of hypertension in both parents before age 60 is cause for exclusion. This exclusion criterion, however, does not apply to discordant sib-pairs.
* Diabetic individuals were excluded. Diabetes uncovered as a result of SAPPHIRe lab work does not lead to exclusion however.
* Severe kidney disease (except stones and remote infections) of creatinine > 1.5 mg/dl, unless documented proof that the subject met inclusion criteria prior to increase in creatinine levels.
* A body-mass index greater than 35.
* In addition, the following conditions are considered as cause for exclusion: ongoing (or within the past 6 months) treatment for cancer; terminal illness (life expectancy fewer than 6 months); liver cirrhosis or any other chronic illness; pregnancy or fewer than 6 months post-partum.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A follow-up genetic study of Taiwan SAPPHIRe Cohort
Sampling Method: Non-Probability Sample
Enrollment: 1246 (Actual)
Dates: Start 2001-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chao Hsiung, PhD, Study Director — Division of Biostatistics and Bioinformatics, National Health Research Institutes
Locations (1):
- Division of Biostatistics and Bioinformatics, NHRI, Miaoli County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee IT, Chiu YF, Hwu CM, He CT, Chiang FT, Lin YC, Assimes T, Curb JD, Sheu WH. Central obesity is important but not essential component of the metabolic syndrome for predicting diabetes mellitus in a hypertensive family-based cohort. Results from the Stanford Asia-pacific program for hypertension and insulin resistance (SAPPHIRe) Taiwan follow-up study. Cardiovasc Diabetol. 2012 Apr 26;11:43. doi: 10.1186/1475-2840-11-43. PMID 22537054